CLINICAL TRIAL: NCT04309006
Title: Volumetric Evaluation of Buccal Soft Tissue Contour Using Customized Healing Abutment During Immediate Implant Placement with Connective Tissue Grafting. a Randomized Controlled Clinical Trial
Brief Title: Buccal Soft Tissue Contour Changes After Immediate Implant Placement with or Without Connective Tissue Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Ahmed Abo El Futtouh, Clinical Director of Implant Program - Periodontology and Implantology Consultant, Misr International University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PER8273003
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Dental Implant Placement
Keywords: Immediate implant placement; Connective tissue graft; buccal soft tissue contour; customized healing abutment; volumetric analysis; cone beam computerized tomography (CBCT)

STUDY DESIGN:
Intervention Model Description: The first factor is the use of connective tissue graft which includes two levels and the second factor is the use of healing abutment which includes two levels.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- CTG and customized healing abutment (Experimental): Customized healing abutment used with connective tissue graft
  Interventions: Procedure: CTG and customized healing abutment
- CTG and conventional healing abutment (Experimental): Conventional healing abutment (same diameter of the implant) used with connective tissue graft
  Interventions: Procedure: CTG and conventional healing abutment
- customized healing abutment (Active Comparator): Customized healing abutment used without connective tissue graft
  Interventions: Procedure: CTG and customized healing abutment
- conventional healing abutment (Active Comparator): Conventional healing abutment (same diameter of the implant) without connective tissue graft
  Interventions: Procedure: CTG and conventional healing abutment

INTERVENTIONS:
Procedure: CTG and customized healing abutment — screw- retained customized healing abutment
  Other Names: zimmer biomed dental implants and connective tissue grafts and customized healing abutments
  Arms: CTG and customized healing abutment; customized healing abutment
Procedure: CTG and conventional healing abutment — conventional healing abutment
  Other Names: Zimmer biomed dental implants and connective tissue graft
  Arms: CTG and conventional healing abutment; conventional healing abutment

SUMMARY:
Statement of the problem: Using customized contoured healing abutments at the time of immediate implant placement is a treatment modality to improve esthetics by maintain the soft tissue contour. Using connective tissue grafts enhances and maintains soft tissue stability. However, the effect of the combined procedures for maintenance of the soft tissue morphology remains unclear. Purpose : The aim of the study is to evaluate the volumetric difference of buccal soft tissue contour around immediate implants placed with and without connective tissue grafts and customized healing abutments. Materials and Methods: Fifty-two patients with single maxillary anterior or premolar tooth indicated for extraction will participate in this study, 13 patients will randomly be assigned in each group. Group 1 (test group) will be treated by immediate implant placement (IIP) with connective tissue graft (CTG) and customized healing abutment, Group 2 (test group) IIP with CTG and healing abutment same diameter of the implant, Group 3 (test group) IIP and customized healing abutment, while the 4th group (control) IIP with healing abutment same diameter of the implant. Extra-oral scanning of the buccal contour will be carried out presurgical and at 3, 6, 9 and 12 months after surgery. Difference in contour gained will be compared to the original contour and between groups. Radiographic evaluation will be done using CBCT at 12 months to measure the bone width. In addition, soft tissue thickness, mid facial recession, gingival biotype, interdental papilla height, soft tissue peri- implant parameters and any surgical or prosthetic complications will be assessed.

DETAILED DESCRIPTION:
After administration of local anaesthesia, the tooth will be extracted by the principle investigator without raising flaps, as atraumatically as possible by using periotomes without disturbing the papillary tissues (minimal traumatic extraction technique). After the extraction of the tooth, the socket will be carefully cleaned to excavate the granulation tissue in the marginal and apical regions. Using standard implant system protocol preparation of the osteotomy will take place. Initial drill will be placed palatally till final drill reached. Placement of the implant without any raising of the flap will be performed in the correct implant position. Primary stability of the implant will be measured by rotational insertion torque value, to be ≥30Ncm (31). After implant placement, the allocation will be revealed to the practitioner for the type of the healing abutment to be used and whether connective tissue graft will be used or not.

Thirteen implants (intervention 1) will receive screw- retained customized healing abutment, and thirteen other implants in the 2nd intervention group will receive the conventional healing abutment of same diameter of the implant. In both groups connective tissue graft will be used. Connective tissue grafts will be harvested from the hard palate and placed at the implant sites in a supraperiosteal partial dissection (pouch technique) prepared at the buccal aspect without using vertical incisions and without flap elevation. Sutures will be used to stabilize the graft in its desired place.

The fabrication of the customized healing abutment is as follows; the temporary cylindrical abutment will be screwed to the implant then flowable composite will be injected at the gingival margin level to adapt to the screw-retained temporary cylindrical abutments that will be sand-blasted for mechanical retention of the composite, taking the shape of the socket at the marginal gingiva. A buccal groove will be made after the polymerization of this material for easier application. The abutments will be removed for final configurations of the apical part mimicking the emergence profile of the extracted tooth and finishing with laboratory discs and burs. The custom healing screw will then be screwed to the implant with the correct torque. Patients will be recalled for regular follow ups. Other thirteen implants (intervention 3) will receive screw- retained customized healing abutment, and for the control (the 4th group) group thirteen implants will receive the conventional healing abutment of same diameter of the implant. No connective tissue grafts are to be used in these two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Adults at or above the age of 18.
2. Patients who have at least one non-restorable maxillary anterior or premolar tooth with sound adjacent teeth.
3. Intact thick biotype gingival tissue with at least 2mm band of keratinized tissue.
4. Buccal bone thickness should be 1mm or less assessed in CBCT with good apical bone.
5. Sagittal root position type 1 as described by Kan et al(24).
6. Good oral hygiene
7. Patient accepts to provide an informed consent

Exclusion Criteria:

1. Smokers
2. Pregnant and lactating females.
3. Medically compromised patients, as Uncontrolled diabetic patients, patients taking bisphosphonates injection for treatment of osteoporosis, patients with active cardiac diseases, patients undergoing radiotherapy or chemotherapy, or any other medical and general contraindications for the surgical procedure (i.e. ASA score ≥III) (25)
4. Patients with active infection related at the site of implant/bone graft placement.
5. Patients with untreated active periodontal diseases.
6. Patients with parafunctional habits.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Volumetric analysis of buccal contour | Before surgery - 3 months - 6 months - 9 months - 12 months
  Measuring changes in the buccal soft tissue contour in comparison to the original ones, at 2,4 and 6 mm from the pre-operative gingival margin. This will be done using Extra oral scanning and 3D viewer software

SECONDARY OUTCOMES:
Bucco-palatal width | Before surgery - 12 months
  Measured using Cone Beam CT
Gingival thickness | Before surgery - 6 months - 12 months
  Measured using Periodontal Probe
Mid facial recession | Before surgery - 3 months - 6 months - 9 months - 12 months
  Measured with 3D viewer software
Interdental papillae height | Before surgery - 3 months - 6 months - 9 months - 12 months
  Measured with 3D viewer software
Modified Plaque Index | 3 months - 6 months - 9 months - 12 months
  Measured with periodontal probe
Modified Bleeding Index | 3 months - 6 months - 9 months - 12 months
  Measured with periodontal probe
Patient satisfaction | 12 months
  Measured with Visual Analogue Scale (VAS) The patients will mark their satisfaction in a non-numerical 100 mm line ranging from "not at all satisfied=0" (left) to "very satisfied=100" (right), for each implant

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed I Abo El Futtouh, Master, Principal Investigator — Clinical Director of Implant Program - Misr International University; Khaled Abdel-Ghaffar, Doctor, Study Director — Minister of Higher Education and Scientific Research; Inas M El-Zayat, Doctor, Study Director — Assoc.Prof - Operative department, Faculty of Dentistry; Mariam S Hanna, Bsc, Study Director — Dentist/Researcher - IDCE; Nael A Mina, Bsc, Study Chair — Misr International University; Abdel Rahman A Abdel Rahman, Master, Study Chair — International Dental Contiuing Education; Ahmed F Mostafa, Bsc, Study Chair — International Dental Contiuing Education
Locations (2):
- Egypt (2):
  - International Dental Contining Education Centre (IDCE), Cairo
  - Misr International University, Cairo

IPD SHARING:
Plan to Share IPD: Yes
All data can be shared
Supporting Information: SAP, CSR
Time Frame: One year
Access Criteria: Principal investigator

REFERENCES:
- [Background] Buser D, Halbritter S, Hart C, Bornstein MM, Grutter L, Chappuis V, Belser UC. Early implant placement with simultaneous guided bone regeneration following single-tooth extraction in the esthetic zone: 12-month results of a prospective study with 20 consecutive patients. J Periodontol. 2009 Jan;80(1):152-62. doi: 10.1902/jop.2009.080360. PMID 19228101
- [Background] Kan JY, Rungcharassaeng K. Site development for anterior single implant esthetics: the dentulous site. Compend Contin Educ Dent. 2001 Mar;22(3):221-6, 228, 230-1; quiz 232. PMID 11913259
- [Background] Fuentealba R, Jofre J. Esthetic failure in implant dentistry. Dent Clin North Am. 2015 Jan;59(1):227-46. doi: 10.1016/j.cden.2014.08.006. Epub 2014 Sep 26. PMID 25434568
- [Background] Goodacre CJ, Kan JY, Rungcharassaeng K. Clinical complications of osseointegrated implants. J Prosthet Dent. 1999 May;81(5):537-52. doi: 10.1016/s0022-3913(99)70208-8. PMID 10220658
- [Background] Kan JY, Rungcharassaeng K, Lozada JL, Zimmerman G. Facial gingival tissue stability following immediate placement and provisionalization of maxillary anterior single implants: a 2- to 8-year follow-up. Int J Oral Maxillofac Implants. 2011 Jan-Feb;26(1):179-87. PMID 21365054
- [Background] Chen ST, Beagle J, Jensen SS, Chiapasco M, Darby I. Consensus statements and recommended clinical procedures regarding surgical techniques. Int J Oral Maxillofac Implants. 2009;24 Suppl:272-8. No abstract available. PMID 19885450
- [Background] De Bruyckere T, Eghbali A, Younes F, De Bruyn H, Cosyn J. Horizontal stability of connective tissue grafts at the buccal aspect of single implants: a 1-year prospective case series. J Clin Periodontol. 2015 Sep;42(9):876-882. doi: 10.1111/jcpe.12448. Epub 2015 Sep 16. PMID 26373422
- [Background] Hammerle CH, Chen ST, Wilson TG Jr. Consensus statements and recommended clinical procedures regarding the placement of implants in extraction sockets. Int J Oral Maxillofac Implants. 2004;19 Suppl:26-8. No abstract available. PMID 15635943
- [Background] Levine RA, Ganeles J, Kan J, Fava PL. 10 Keys for Successful Esthetic-Zone Single Implants: Importance of Biotype Conversion for Lasting Success. Compend Contin Educ Dent. 2018 Sep;39(8):522-529; quiz 530. PMID 30188147
- [Background] Lee CT, Tao CY, Stoupel J. The Effect of Subepithelial Connective Tissue Graft Placement on Esthetic Outcomes After Immediate Implant Placement: Systematic Review. J Periodontol. 2016 Feb;87(2):156-67. doi: 10.1902/jop.2015.150383. Epub 2015 Oct 15. PMID 26469808
- [Background] Kolerman R, Nissan J, Mijiritsky E, Hamoudi N, Mangano C, Tal H. Esthetic assessment of immediately restored implants combined with GBR and free connective tissue graft. Clin Oral Implants Res. 2016 Nov;27(11):1414-1422. doi: 10.1111/clr.12755. Epub 2016 Jan 7. PMID 26743894
- [Background] Cosyn J, Eghbali A, Hermans A, Vervaeke S, De Bruyn H, Cleymaet R. A 5-year prospective study on single immediate implants in the aesthetic zone. J Clin Periodontol. 2016 Aug;43(8):702-9. doi: 10.1111/jcpe.12571. Epub 2016 Jun 13. PMID 27120578
- [Background] Touati B, Guez G, Saadoun A. Aesthetic soft tissue integration and optimized emergence profile: provisionalization and customized impression coping. Pract Periodontics Aesthet Dent. 1999 Apr;11(3):305-14; quiz 316. PMID 10379291
- [Background] Saito H, Chu SJ, Reynolds MA, Tarnow DP. Provisional Restorations Used in Immediate Implant Placement Provide a Platform to Promote Peri-implant Soft Tissue Healing: A Pilot Study. Int J Periodontics Restorative Dent. 2016 Jan-Feb;36(1):47-52. doi: 10.11607/prd.1945. PMID 26697547
- [Background] del Castillo RA. Immediate provisionalization of a single-tooth implant with a temporary cylinder in one surgical appointment. Pract Proced Aesthet Dent. 2006 Jun;18(5):suppl 3-5. No abstract available. PMID 16903535
- [Background] Lemongello GJ Jr. Immediate custom implant provisionalization: a prosthetic technique. Pract Proced Aesthet Dent. 2007 Jun;19(5):273-9. PMID 17679316
- [Background] Mihali S. Maintaining Tissue Architecture in Immediate Implant Placement Following Extraction of Natural Teeth Using Custom Healing Screw. Biomed J Sci Tech Res. 2018
- [Background] Akin R. A New Concept in Maintaining the Emergence Profile in Immediate Posterior Implant Placement: The Anatomic Harmony Abutment. J Oral Maxillofac Surg. 2016 Dec;74(12):2385-2392. doi: 10.1016/j.joms.2016.06.184. Epub 2016 Jul 1. PMID 27475245
- [Background] Janakievski J. Case Report : Maintenance of Gingival Form Following Immediate Implant Placement - The Custom-Healing Abutment. Adv Esthet Interdiscip Dent. 2007;3(4):4-7
- [Background] Kan JYK, Rungcharassaeng K, Deflorian M, Weinstein T, Wang HL, Testori T. Immediate implant placement and provisionalization of maxillary anterior single implants. Periodontol 2000. 2018 Jun;77(1):197-212. doi: 10.1111/prd.12212. Epub 2018 Feb 25. PMID 29478284
- [Background] van Nimwegen WG, Raghoebar GM, Zuiderveld EG, Jung RE, Meijer HJA, Muhlemann S. Immediate placement and provisionalization of implants in the aesthetic zone with or without a connective tissue graft: A 1-year randomized controlled trial and volumetric study. Clin Oral Implants Res. 2018 Jul;29(7):671-678. doi: 10.1111/clr.13258. Epub 2018 May 27. PMID 29806181
- [Background] Luckerath W, Roder L, Enkling N. The Effect of Primary Stabilization of the Graft in a Combined Surgical and Prosthodontic Ridge Preservation Protocol: A Prospective Controlled Clinical Pilot Study. Int J Periodontics Restorative Dent. 2018 May/Jun;38(3):e49-e58. doi: 10.11607/prd.3172. PMID 29641631
- [Background] Kan JY, Roe P, Rungcharassaeng K, Patel RD, Waki T, Lozada JL, Zimmerman G. Classification of sagittal root position in relation to the anterior maxillary osseous housing for immediate implant placement: a cone beam computed tomography study. Int J Oral Maxillofac Implants. 2011 Jul-Aug;26(4):873-6. PMID 21841998
- [Background] Smeets EC, de Jong KJ, Abraham-Inpijn L. Detecting the medically compromised patient in dentistry by means of the medical risk-related history. A survey of 29,424 dental patients in The Netherlands. Prev Med. 1998 Jul-Aug;27(4):530-5. doi: 10.1006/pmed.1998.0285. PMID 9672946
- [Background] Chrcanovic BR, Kisch J, Albrektsson T, Wennerberg A. Factors Influencing Early Dental Implant Failures. J Dent Res. 2016 Aug;95(9):995-1002. doi: 10.1177/0022034516646098. Epub 2016 May 4. PMID 27146701
- [Background] Olmedo-Gaya MV, Manzano-Moreno FJ, Canaveral-Cavero E, de Dios Luna-del Castillo J, Vallecillo-Capilla M. Risk factors associated with early implant failure: A 5-year retrospective clinical study. J Prosthet Dent. 2016 Feb;115(2):150-5. doi: 10.1016/j.prosdent.2015.07.020. Epub 2015 Nov 3. PMID 26545864
- [Background] Vissink A, Spijkervet F, Raghoebar GM. The medically compromised patient: Are dental implants a feasible option? Oral Dis. 2018 Mar;24(1-2):253-260. doi: 10.1111/odi.12762. PMID 29480621
- [Background] Lobbezoo F, Brouwers JE, Cune MS, Naeije M. Dental implants in patients with bruxing habits. J Oral Rehabil. 2006 Feb;33(2):152-9. doi: 10.1111/j.1365-2842.2006.01542.x. PMID 16457676
- [Background] Kan JY, Morimoto T, Rungcharassaeng K, Roe P, Smith DH. Gingival biotype assessment in the esthetic zone: visual versus direct measurement. Int J Periodontics Restorative Dent. 2010 Jun;30(3):237-43. PMID 20386780
- [Background] Testori T, Meltzer A, Del Fabbro M, Zuffetti F, Troiano M, Francetti L, Weinstein RL. Immediate occlusal loading of Osseotite implants in the lower edentulous jaw. A multicenter prospective study. Clin Oral Implants Res. 2004 Jun;15(3):278-84. doi: 10.1111/j.1600-0501.2004.01013.x. PMID 15142089
- [Background] Araujo MG, Lindhe J. Dimensional ridge alterations following tooth extraction. An experimental study in the dog. J Clin Periodontol. 2005 Feb;32(2):212-8. doi: 10.1111/j.1600-051X.2005.00642.x. PMID 15691354
- [Background] Zuhr O, Baumer D, Hurzeler M. The addition of soft tissue replacement grafts in plastic periodontal and implant surgery: critical elements in design and execution. J Clin Periodontol. 2014 Apr;41 Suppl 15:S123-42. doi: 10.1111/jcpe.12185. PMID 24640997
- [Background] Ueno D, Kobayashi M, Tanaka K, Watanabe T, Nakamura T, Ueda K, Nagano T. Measurement accuracy of alveolar soft tissue contour using a laboratory laser scanner. Odontology. 2018 Apr;106(2):202-207. doi: 10.1007/s10266-017-0315-4. Epub 2017 Aug 2. PMID 28770415
- [Background] Kim SH, Choi JH, Chung KR, Nelson G. Do sand blasted with large grit and acid etched surface treated mini-implants remain stationary under orthodontic forces? Angle Orthod. 2012 Mar;82(2):304-12. doi: 10.2319/032511-212.1. Epub 2011 Aug 10. PMID 21830933
- [Background] Koerich L, Weissheimer A, Koerich LE, Luz D, Deeb JG. A Technique of Cone-Beam Computerized Tomography Superimposition in Implant Dentistry. J Oral Implantol. 2018 Oct;44(5):365-369. doi: 10.1563/aaid-joi-D-17-00282. Epub 2018 May 2. No abstract available. PMID 29717909
- [Background] Amid R, Mirakhori M, Safi Y, Kadkhodazadeh M, Namdari M. Assessment of gingival biotype and facial hard/soft tissue dimensions in the maxillary anterior teeth region using cone beam computed tomography. Arch Oral Biol. 2017 Jul;79:1-6. doi: 10.1016/j.archoralbio.2017.02.021. Epub 2017 Mar 1. PMID 28279824
- [Background] Cevidanes LH, Styner MA, Proffit WR. Image analysis and superimposition of 3-dimensional cone-beam computed tomography models. Am J Orthod Dentofacial Orthop. 2006 May;129(5):611-8. doi: 10.1016/j.ajodo.2005.12.008. PMID 16679201
- [Background] Borges GJ, Ruiz LF, de Alencar AH, Porto OC, Estrela C. Cone-beam computed tomography as a diagnostic method for determination of gingival thickness and distance between gingival margin and bone crest. ScientificWorldJournal. 2015;2015:142108. doi: 10.1155/2015/142108. Epub 2015 Mar 31. PMID 25918737
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627